CLINICAL TRIAL: NCT01094652
Title: The Addition of Whole Grains to the Diets of Middle-school Children: A Study of Digestive Health and Immune Defenses
Brief Title: The Addition of Whole Grains to the Diets of Middle-school Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: University of Florida (Other)
Collaborators: General Mills (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Basic Science
Other Study IDs: 480-2009
Record Dates: First submitted 2010-03-23; First posted 2010-03-29 (Estimated); Last update posted 2012-08-02 (Estimated); Status verified 2012-07

CONDITIONS: Healthy
Keywords: Adolescent; Whole grain; Digestive health; Dietary fiber; Grain; Microbiota; Inflammation; Mucosal Immunity
MeSH Terms: conditions — Inflammation

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Whole grain diet (Experimental): Participants in this group will be given whole grain snacks on school days and food packages consisting of whole grain breads, breakfast cereals, rice, snack foods, and pasta to replace their typical grains consumed at home.
  Interventions: Dietary Supplement: Whole grain diet
- Refined grain diet (Active Comparator): Participants in this group will be given refined grain snacks on school days and food packages consisting of refined grain breads, breakfast cereals, rice, snack foods, and pasta to replace their typical grains consumed at home.
  Interventions: Dietary Supplement: Refined grain diet

INTERVENTIONS:
Dietary Supplement: Whole grain diet — Subjects were told to consume three different kinds of study food each day. The goal was an intake of greater than or equal to 80 g of whole grains per day.
  Arms: Whole grain diet
Dietary Supplement: Refined grain diet — The refined grain food products were matched as closely as possible to the foods contained in the whole grain diet. Subjects were told to consume three different kinds of study food each day.
  Arms: Refined grain diet

SUMMARY:
The Dietary Guidelines for Americans recommend that children and adolescents "consume whole-grain products often; at least half the grains should be whole grains." Few, if any studies, examine the benefit of whole grains on the health of adolescents. The purpose of this study is to determine if adolescents eating diets rich in whole grains vs. diets rich in refined grains (i.e., a typical diet) have improved markers of digestive and immune health.

DETAILED DESCRIPTION:
Middle-school students will be recruited and randomized to receive >/=80 g of whole grains (>/=5 servings) or similar foods made with refined grains each day for six weeks. Based on treatment group, subjects will be provided either whole grain or refined grain foods and snacks. They will be instructed on how to use these foods to replace other foods already contained in the diet. Stool, blood, and saliva samples will be obtained at baseline and at study end to examine the microbiota and markers of digestive and immune health. Daily records will be maintained by the students to assess bowel habits and compliance. It is anticipated that whole grains will increase stool bulk resulting in increased stool frequency and softer stools. Additionally, fermentation of the fiber within the colon will alter the microbiota profile. Because the majority of the immune system resides within the gastrointestinal tract, improved balance of the intestinal microbiota may prime the immune system thus contributing to improved immune defense.

ELIGIBILITY:
Inclusion Criteria:

* Middle-school student at Westwood Middle School, Gainesville, FL
* Parental/guardian consent
* Willing to eat three different study foods each day for six weeks
* Willing to provide two blood samples and two saliva samples over the course of the study

Exclusion Criteria:

* Taking medications for constipation or diarrhea
* Antibiotic therapy within the past four weeks prior to randomization
* Takes probiotics or consumes greater than three servings of yogurt per week
* Has any diseases or illnesses such as gastrointestinal disease (gastric ulcers, Crohn's, ulcerative colitis, etc.), other chronic diseases (diabetes, kidney disease, etc.) or immune-modulating diseases (HIV, AIDS, autoimmune, hepatitis, cancer, etc.)
* Has any food allergies (wheat, soy, egg, milk, gluten, nuts, or any other food or food ingredient)

Ages: 11 Years to 15 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child
Enrollment: 83 (Actual)
Dates: Start 2010-02; Primary Completion 2010-04 (Actual); Study Completion 2010-04 (Actual)

PRIMARY OUTCOMES:
Stool frequency | 6 weeks

SECONDARY OUTCOMES:
Changes in overall microbiota diversity | 6 weeks
  Microbial diversity will be measured by DGGE profiling to detect large distortions. Quantitative changes in the proportions of select bacteria will be measured using qPCR.
Inflammatory markers | 6 weeks
  Serum CRP, fibrinogen, IL-1, IL-6, and antioxidant capacity; mitogen-induced cytokine production including Th1, Th2, and inflammatory cytokines
Secretory IgA | 6 weeks
  Salivary and fecal sIgA

CONTACTS AND LOCATIONS:
Overall Officials: Bobbi Langkamp-Henken, PhD, RD, Principal Investigator — University of Florida
Locations (1):
- Westwood Middle School, Gainesville, Florida, United States

REFERENCES:
- [Derived] Langkamp-Henken B, Nieves C Jr, Culpepper T, Radford A, Girard SA, Hughes C, Christman MC, Mai V, Dahl WJ, Boileau T, Jonnalagadda SS, Thielecke F. Fecal lactic acid bacteria increased in adolescents randomized to whole-grain but not refined-grain foods, whereas inflammatory cytokine production decreased equally with both interventions. J Nutr. 2012 Nov;142(11):2025-32. doi: 10.3945/jn.112.164996. Epub 2012 Sep 26. PMID 23014489